CLINICAL TRIAL: NCT03790592
Title: Visual Outcomes and Patient Satisfaction After Presbyopic Lens Exchange With a Trifocal Intraocular Lens (IOL)
Brief Title: Visual Outcomes After Presbyopic Lens Exchange
Acronym: RELAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LISA tri 839MP BER-401-18
Record Dates: First submitted 2018-12-28; First posted 2018-12-31 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- trifocal IOL (Experimental): patients implanted with a trifocal intraocular lens
  Interventions: Device: trifocal IOL

INTERVENTIONS:
Device: trifocal IOL — intraocular lens

SUMMARY:
Evaluation of mean preoperative and postoperative Corrected distance visual acuity (CDVA) after Refractive Lens Exchange in presbyopic patients

DETAILED DESCRIPTION:
Compare preoperative and postoperative Corrected distance visual acuity

ELIGIBILITY:
Inclusion Criteria:

1. Patient informed of the consequences and constraints of the protocol and who has given his/her written informed consent
2. Patients of any gender, aged 18 years or older
3. Assured follow-up examinations
4. Post-operative astigmatism ≤ 0.75 Diopter
5. IOL implanted into the capsular bag with trifocal IOL in both eyes
6. Patients who had bilateral uncomplicated presbyopic lens exchange surgery in both healthy eyes
7. Preoperative monocular and binocular CDVA equal or better than 0.2 logMAR
8. Normal findings in the medical history and physical examination

Exclusion Criteria:

1. Patients unable to meet the limitations of the protocol or likely of non-cooperation during the trial
2. Patients whose freedom is impaired by administrative or legal order
3. Concurrent participation in another drug or device investigation that affects patients vision
4. Signs of early cataract in either eye
5. Preoperative monocular and binocular CDVA worse than 0.2 logMAR
6. Clinically significant Posterior capsule opacification (PCO) defined as a CDVA loss of 0.2 logMAR or more in either eye
7. Cataract of any grade
8. Ocular disorders, that could potentially cause future acuity loss to a level of 0.20 logMAR (best-corrected) or worse in either eye
9. Any anterior segment pathology that could significantly affect outcomes (e.g. chronic uveitis, iritis, aniridia, rubeosis iridis, clinically significant anterior membrane dystrophies, poor pupil dilation, etc.)
10. Abnormal corneal findings in either eye (e.g. keratoconus, pellucid marginal degeneration, or irregular astigmatism, clinically significant corneal membrane dystrophies)
11. Any condition in the study eye that could affect IOL stability (e.g. zonular dialysis, evident zonular weakness or dehiscence, etc.)
12. History of any clinically significant retinal pathology or ocular diagnosis (e.g. diabetic retinopathy, ischemic diseases, macular degeneration, retinal detachment, optic neuropathy optic nerv atrophy, amblyopia, strabismus, microphthalmos, aniridia, epiretinal membrane etc.) in the study eyes that could alter or limit final postoperative visual prognosis.
13. Patients, who are unable to fixate for a longer time, e.g. strabismus, nystagmus
14. Patient expected to require retinal laser treatment before 6 month follow-up visit
15. Patient require refractive laser treatment / refractive laser touch-up before 6 month follow up visit
16. Current Systemic or ocular pharmacotherapy that effects patients vision
17. Floppy iris syndrome
18. Monophthalmic patient
19. Previous corneal surgery
20. Previous use of cytotoxic drugs or total body irradiation
21. Dementia
22. Uncontrolled glaucoma or Intraocular pressure (IOP) higher than 24 millimeter of mercury (mmHg) under ocular hypertension treatment
23. Any other pathology or condition presenting, according to the investigator opinion, a risk for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Corrected distance visual acuity | 4 to 6 months postop
  preoperative and postoperative Corrected distance visual acuity will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Augenzentrum Michelfeld, Michelfeld, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez J, Alfonso Sanchez JF, Nieradzik M, Valcarcel B, Burguera N, Kapp A. Visual performance, safety and patient satisfaction after bilateral implantation of a trifocal intraocular lens in presbyopic patients without cataract. BMC Ophthalmol. 2022 Aug 10;22(1):341. doi: 10.1186/s12886-022-02556-y. PMID 35948879